CLINICAL TRIAL: NCT02557204
Title: Comparison of Different Methods of Nasogastric Tube Insertion in Anesthetized and Intubated Patients: A Prospective Randomized Controlled Trial
Brief Title: Comparison of Different Methods of Nasogastric Tube Insertion in Anesthetized and Intubated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AntalyaTRH 007
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Disorder of Abdomen
Keywords: nasogastric tube insertion; Video laryngoscope; success rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- conventional technique (Active Comparator): the nasogastric tube will be inserted gently through a selected nostril with the head being maintained in the neutral position.
  Interventions: Procedure: conventional technique
- head in the lateral position technique (Experimental): the patient's head will be turned to the right lateral position. Nasogastric tube will be inserted through the right nostril without any maneuvers of the neck.
  Interventions: Procedure: head in the lateral position technique
- endotracheal tube assisted technique (Experimental): Nasogastric tube will be inserted the trimmed 7.5 mm internal diameter endotracheal tube what cut proximal end with sterile scissors and endotracheal tube will be advanced blindly into the oral cavity to a depth of approximately 18 cm without laryngoscope together the nasogastric tube.
  Interventions: Procedure: endotracheal tube assisted technique
- videolaryngoscope technique (Experimental): Nasogastric tube was inserted transnasally and advanced into esophagus under direct vision.
  Interventions: Procedure: videolaryngoscope technique

INTERVENTIONS:
Procedure: conventional technique — the nasogastric tube will be inserted gently through a selected nostril with the head being maintained in the neutral position.
  Arms: conventional technique
Procedure: head in the lateral position technique — the patient's head will be turned to the right lateral position. Nasogastric tube will be inserted through the right nostril without any maneuvers of the neck.
  Arms: head in the lateral position technique
Procedure: endotracheal tube assisted technique — Nasogastric tube will be inserted the trimmed 7.5 mm internal diameter endotracheal tube what cut proximal end with sterile scissors and endotracheal tube will be advanced blindly into the oral cavity to a depth of approximately 18 cm without laryngoscope together the nasogastric tube.
  Arms: endotracheal tube assisted technique
Procedure: videolaryngoscope technique — Nasogastric tube was inserted transnasally and advanced into esophagus under direct vision.
  Arms: videolaryngoscope technique

SUMMARY:
The primary aim of this study is to investigate the difference in the first attempt and overall success rate of different techniques for insertion of nasogastric tube. Secondary aim is to investigate the difference of the duration of insertion using the selected technique, complications during insertion such as kinking, knotting, mucosal bleeding

DETAILED DESCRIPTION:
Two hundred adult patients, who received general anaesthesia for elective abdominal surgeries that required nasogastric tube insertion, will be randomized by means of a computer-generated randomization order into four groups: Conventional group (Group C), head in the lateral position group (Group L), endotracheal tube assisted group (group ET) and video laryngoscope group (group MG).

Success rate of the selected technique (first attempt, second attempt and overall), duration of insertion for selected technique, complications such as kinking and mucosal bleeding will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received general anaesthesia for elective abdominal surgeries that required nasogastric tube insertion.

Exclusion Criteria:

* Patients with a history of coagulopathy,
* nasal stenosis,
* upper respiratory tract diseases or anomalies,
* esophageal varix, esophageal hiatus hernia,
* base of skull fracture,
* loose teeth,
* Cormack and Lehane and/or Mallampati scores of 3 or 4,
* patients younger than 18 years and older than 70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
difference in the first attempt and overall success rate | participants will be followed to the starting from the NG tube insert through the nostril until the confirm to successful insertion into stomach.
  investigate the difference in the first attempt and overall success rate (with percentage) of different techniques for insertion of nasogastric tube.

SECONDARY OUTCOMES:
difference of the duration of insertion and complications during insertion | participants will be followed for the duration of intraoperative period and postoperative 4 hours.
  investigate the difference of the duration of insertion (in seconds) using the selected technique and complications (with number and percentage) during insertion such as kinking, knotting, mucosal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ali S Kavakli, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Kirtania J, Ghose T, Garai D, Ray S. Esophageal guidewire-assisted nasogastric tube insertion in anesthetized and intubated patients: a prospective randomized controlled study. Anesth Analg. 2012 Feb;114(2):343-8. doi: 10.1213/ANE.0b013e31823be0a4. Epub 2011 Nov 21. PMID 22104075
- [Background] Moharari RS, Fallah AH, Khajavi MR, Khashayar P, Lakeh MM, Najafi A. The GlideScope facilitates nasogastric tube insertion: a randomized clinical trial. Anesth Analg. 2010 Jan 1;110(1):115-8. doi: 10.1213/ANE.0b013e3181be0e43. Epub 2009 Oct 27. PMID 19861362
- [Background] Appukutty J, Shroff PP. Nasogastric tube insertion using different techniques in anesthetized patients: a prospective, randomized study. Anesth Analg. 2009 Sep;109(3):832-5. doi: 10.1213/ane.0b013e3181af5e1f. PMID 19690254
- [Background] Kwon OS, Cho GC, Jo CH, Cho YS. Endotracheal tube-assisted orogastric tube insertion in intubated patients in an ED. Am J Emerg Med. 2015 Feb;33(2):177-80. doi: 10.1016/j.ajem.2014.11.004. Epub 2014 Nov 13. PMID 25435406
- [Background] Chun DH, Kim NY, Shin YS, Kim SH. A randomized, clinical trial of frozen versus standard nasogastric tube placement. World J Surg. 2009 Sep;33(9):1789-92. doi: 10.1007/s00268-009-0144-x. PMID 19626360
- [Background] Bong CL, Macachor JD, Hwang NC. Insertion of the nasogastric tube made easy. Anesthesiology. 2004 Jul;101(1):266. doi: 10.1097/00000542-200407000-00058. No abstract available. PMID 15220819
- [Background] Ghatak T, Samanta S, Baronia AK. A new technique to insert nasogastric tube in an unconscious intubated patient. N Am J Med Sci. 2013 Jan;5(1):68-70. doi: 10.4103/1947-2714.106215. PMID 23378961
- [Background] Tsai YF, Luo CF, Illias A, Lin CC, Yu HP. Nasogastric tube insertion in anesthetized and intubated patients: a new and reliable method. BMC Gastroenterol. 2012 Aug 1;12:99. doi: 10.1186/1471-230X-12-99. PMID 22853453
- [Background] Okabe T, Goto G, Hori Y, Sakamoto A. Gastric tube insertion under direct vision using the King Vision video laryngoscope: a randomized, prospective, clinical trial. BMC Anesthesiol. 2014 Sep 25;14:82. doi: 10.1186/1471-2253-14-82. eCollection 2014. PMID 25278810
- [Background] Illias AM, Hui YL, Lin CC, Chang CJ, Yu HP. A comparison of nasogastric tube insertion techniques without using other instruments in anesthetized and intubated patients. Ann Saudi Med. 2013 Sep-Oct;33(5):476-81. doi: 10.5144/0256-4947.2013.476. PMID 24188942
- [Background] Milsom SA, Sweeting JA, Sheahan H, Haemmerle E, Windsor JA. Naso-enteric Tube Placement: A Review of Methods to Confirm Tip Location, Global Applicability and Requirements. World J Surg. 2015 Sep;39(9):2243-52. doi: 10.1007/s00268-015-3077-6. PMID 25900711
- [Background] Halloran O, Grecu B, Sinha A. Methods and complications of nasoenteral intubation. JPEN J Parenter Enteral Nutr. 2011 Jan;35(1):61-6. doi: 10.1177/0148607110370976. Epub 2010 Oct 26. PMID 20978245